CLINICAL TRIAL: NCT04385251
Title: An International Observational Study of Outpatients With SARS-CoV-2 Infection
Brief Title: International SARS-CoV-2 (COVID-19) Infection Observational Study
Acronym: ICOS
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: ICOS; 75N91019D00024 (Other Grant/Funding Number: Leidos Biomedical Research, Inc.)
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: COVID; COVID19; SARS-CoV 2; Dyspnea
MeSH Terms: conditions — COVID-19; Dyspnea | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At the time of enrollment, selected sites participating in a sub-study will be asked to obtain separate consents for 1) an upper respiratory swab and a blood sample sufficient for four 1mL transport tubes of serum to be shipped to a central repository for future research on COVID-19; and 2) co-enrollment in the INSIGHT Genomics Study (INSIGHT 004) where a blood sample sufficient for six 1mL aliquots of whole blood will be collected. These specimens will be sent to a central repository in the United States for storage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SARS-CoV-2 infection/COVID-19: Adults who present for SARS-CoV-2 testing will be consented for this study. Participants who are enrolled will be informed that if they have SARS-CoV-2 infection/COVID-19, they will be followed for 28 days in an observational cohort study, and that if they do not have SARS-CoV-2 infection, there will be no further follow-up.
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — DATA COLLECTION AT ENROLLMENT:
  Demographics; Symptoms and health status; Co-morbidities; Targeted medications; Specimen Collection (substudy at selected sites): Upper respiratory swab, blood for serum storage.
  DATA COLLECTION AT DAYS 7, 14 & 28:
  Vital and hospitalization status; Symptoms and health status

SUMMARY:
The general aim of this study is to estimate the rate of disease progression for adults testing positive for SARS-CoV-2. The primary endpoint for this study and the basis for sample size is hospitalization or death during the 28 day follow-up period. In some locations special facilities are being built/utilized for quarantine/public health reasons for those who are SARS-CoV-2 positive. Hospitalization is defined as a stay for at least 18 hours, irrespective of reason, at a hospital or one of these special facilities after study enrollment.

Secondary outcomes include participant-reported health status and change in severity of dyspnoea.

DETAILED DESCRIPTION:
SARS-CoV-2 is a coronavirus that emerged in China in late 2019 causing a novel Corona-Virus Induced Disease (COVID-19). COVID-19 is spreading rapidly throughout the world. While a proportion of people with COVID-19 have sufficiently severe symptoms to require hospitalization at the time of initial symptom onset, in others the disease may remain mild, and in some cases there has been observed a worsening of symptoms a few days after initial presentation with relatively mild symptoms. There is an urgent need for understanding the progression of disease for individuals with SARS-CoV-2 infection/COVID-19 who do not require immediate hospitalization.

This is an international, observational cohort study of adults with SARS-CoV-2 infection/COVID-19 managed as outpatients (not hospitalized). This study will also be a platform for the enrollment of outpatients for randomized trials that will be conducted by the INSIGHT group.

Those with confirmed SARS-CoV-2 infection will form an observational cohort study and be followed for 28 days. Procedures and data collection have been streamlined to facilitate the enrollment of a large number of adults at INSIGHT sites around the world.

ELIGIBILITY:
Inclusion Criteria:

- Not currently hospitalized

Exclusion Criteria:

- Persons with a known positive SARS-CoV-2 test > 28 days ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who test positive for SARS-CoV-2 infection/COVID-19 will be followed for 28 days in an observational cohort study.
Sampling Method: Probability Sample
Enrollment: 11973 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Time to Hospitalization | 28 days
  Outcome reported as the mean number of days from enrollment to hospitalization due to COVID-19.
Time to Expiration | 28 days
  Outcome reported as the mean number of days from enrollment to expiration (death) due to COVID-19.

SECONDARY OUTCOMES:
Rate of Death at 7 Days | 7 days
  Outcome reported as the percent of participants who expire due to COVID-19 at 7 days post enrollment.
Rate of Death at 14 Days | 14 days
  Outcome reported as the percent of participants who expire due to COVID-19 at 14 days post enrollment.
Rate of Death at 28 Days | 28 days
  Outcome reported as the percent of participants who expire due to COVID-19 at 28 days post enrollment.
Rate of Hospitalization at 7 Days | 7 days
  Outcome reported as the percent of participants who are hospitalized due to COVID-19 at 7 days post enrollment.
Rate of Hospitalization at 14 Days | 14 days
  Outcome reported as the percent of participants who are hospitalized due to COVID-19 at 14 days post enrollment.
Rate of Hospitalization at 28 Days | 28 days
  Outcome reported as the percent of participants who are hospitalized due to COVID-19 at 28 days post enrollment.
Participant Health at 7 Days | 7 days
  Outcome reported as the percent of participants who are in excellent or very good health at 7 days post enrollment.
Participant Health at 14 Days | 14 days
  Outcome reported as the percent of participants who are in excellent or very good health at 14 days post enrollment.
Participant Health at 28 Days | 28 days
  Outcome reported as the percent of participants who are in excellent or very good health at 28 days post enrollment.
Modified Borg Dyspnea Scale at 7 Days | 7 Days
  The Modified Borg Dyspnea scale (MBDS) contains 12 numeric values which designate the severity of dyspnea symptoms (0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10). Higher scores indicate greater dyspnea severity. Outcome is reported as the mean MBDS score at 7 days post enrollment.
Modified Borg Dyspnea Scale at 14 Days | 14 Days
  The Modified Borg Dyspnea scale (MBDS) contains 12 numeric values which designate the severity of dyspnea symptoms (0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10). Higher scores indicate greater dyspnea severity. Outcome is reported as the mean MBDS score at 14 days post enrollment.
Modified Borg Dyspnea Scale at 28 Days | 28 Days
  The Modified Borg Dyspnea scale (MBDS) contains 12 numeric values which designate the severity of dyspnea symptoms (0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10). Higher scores indicate greater dyspnea severity. Outcome is reported as the mean MBDS score at 28 days post enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: James Neaton, PhD, Principal Investigator — University of Minnesota
Locations (4):
- Denver Public Health, Denver, Colorado, United States
- Hospital General de Agudos JM Ramos Mejia Servicio de Inmunocomprometidos, Buenos Aires, Argentina
- CHIP Department of Infectious Diseases, Copenhagen, Denmark
- University College London Medical School Centre for Sexual Health and HIV Research, London, England, United Kingdom

DOCUMENTS (2):
  • Study Protocol (2020-08-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT04385251/Prot_000.pdf
  • Informed Consent Form (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT04385251/ICF_001.pdf